CLINICAL TRIAL: NCT06499519
Title: Clinical Diagnostic Performance of the SpinChip High-sensitivity Cardiac Troponin I (SpinChip Hs-cTnI) Test
Brief Title: SpinChip Hs-cTnI Clinical Diagnostic Performance
Acronym: HEAT-4
Status: Completed | Type: Observational
Sponsor: SpinChip Diagnostics ASA (Industry)
Collaborators: Aurevia (Industry)
Responsible Party: Sponsor
Other Study IDs: Design Protocol-02856; CIV-23-12-045095 (Other: EUDAMED)
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; High-sensitive; Point of Care; Troponin I; Near-patient test; Heart attack; Diagnostic accuracy
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Li-heparin plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SpinChip hs-cTnI — SpinChip Platform, consisting of the SpinChip hs-cTnI test (self-contained cartridge) and SpinChip Analyzer (instrument)

SUMMARY:
During a heart attack, the protein troponin I is released from the heart muscle into the bloodstream. Measurements of cardiac troponin in blood are used as an aid in the diagnosis of heart attack. The SpinChip hs-cTnI test is a new high-sensitive test for measuring the amount of cardiac troponin I in the bloodstream as an aid in the diagnosis of heart attack.

The purpose of this study is to evaluate the diagnostic accuracy and safety of the SpinChip hs-cTnI test relative to a clinically validated hs-cTnI method.

DETAILED DESCRIPTION:
Cardiac troponins are widely used as a biomarker to aid in the diagnosis of acute myocardial infarction (AMI). These structural proteins are essential in regulating contraction in cardiac muscle cells, and they are sensitive and specific biochemical markers of myocardial damage.

During a heart attack, cardiac muscle cells are injured and release the cardiac marker troponin I (cTnI) into the bloodstream. High-sensitive troponin tests may detect the increase of cardiac troponin in blood within hours after the symptoms of a heart attack has started.

The SpinChip high-sensitivity cardiac troponin I (hs-cTnI) test is a new high-sensitive test for measuring troponin I in blood samples, and the analysis may be performed close to the patient (near-patient test). The results may be obtained within 10 minutes, compared to approximately 1 hour for normal laboratory analysis.

The SpinChip Platform consists of the SpinChip hs-cTnI test and the SpinChip Analyzer and may be used at the emergency department to evaluate patients presenting with symptoms of acute myocardial infarction (chest pain). The test can use blood from finger prick or venous blood samples, either as whole blood or separated into plasma

This study is a multicentre, prospective, observational, non-randomised, open clinical performance study for evaluation of the diagnostic accuracy and safety of the SpinChip hs-cTnI test as an aid in the diagnosis of AMI. Subjects presenting with acute chest discomfort or other symptoms suggestive of AMI will be recruited at the emergency departments (EDs).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed written informed consent
* Subjects ≥ 18 years old
* Subjects presenting at the ED with acute chest discomfort including "pain", "pressure", "tightness", "burning", or "stabbing" and/or other symptoms suggestive of AMI such as upper abdominal pain, left shoulder/arm pain, pain in the jaw, or pain between the scapulae.

Exclusion Criteria:

* Subjects experiencing shock
* Self-reported pregnancy
* Previously included in the study (e.g., in case of a second presentation)
* Patient incapable of judgement, for example due to severe pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to the emergency department with acute chest discomfort or other symptoms suggestive of AMI. This multicentre study will be conducted at up to 10 sites in the EU/EEA, Switzerland and UK.
Sampling Method: Non-Probability Sample
Enrollment: 1551 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristics (AUROC) curve for cTnI concentrations measured at admission to the emergency department (ED) | Day of admission
  Calculate and compare the area under the curve (AUC) for both SpinChip hs-cTnI and clinically validated hs-cTnI method using centrally adjudicated diagnosis of AMI

SECONDARY OUTCOMES:
AUROC for cTnI concentrations measured at 1, 2 and 3 hours after admission to the ED | Day of admission
  Calculate and compare the area under the curve (AUC) for both SpinChip hs-cTnI and clinically validated hs-cTnI method using centrally adjudicated diagnosis of AMI for the given timepoints
Negative predictive value (NPV) at 0, 1, 2, and 3 hours after admission to the ED using the 99th percentile upper reference limit as clinical cut-off | Day of admission
  NPV is defined as the proportion of subjects with measured cTnI concentrations below a clinical cut-off value, who are correctly diagnosed as not having MI.
  The NPVs of the SpinChip hs-cTnI test will be calculated for 0, 1, 2, and 3 hours timepoints, using the overall and sex-specific 99th percentile upper reference limits as clinical cut-offs.
Positive predictive value (PPV) at 0, 1, 2, and 3 hours after admission to the ED using the 99th percentile upper reference limit as clinical cut-off | Day of admission
  PPV is defined as the proportion of subjects with measured cTnI concentrations above a clinical cut-off value, who are diagnosed with MI.
  The PPV of the SpinChip hs-cTnI test will be calculated for cTnI concentrations obtained 0, 1, 2, and 3 hours timepoints, using the overall and sex-specific 99th percentile URL as clinical cut-offs.
Occurrence of MI and/or cardiovascular death (CV) within 30 days | 30 days
  Prognostic accuracy for risk of MI/CV death for 30 days evaluated using Kaplan-Meier plots
  Cox proportional hazard model will be used to evaluate the prognostic performance of the SpinChip hs-cTnI test for outcomes MI and CV death within 30 days.
Derivation and validation of rule-in/rule-out 0/1h and 0/2h algorithms | Day of admission
  Rule-in/rule-out algorithms will be calculated in accordance with the European Society of Cardiology (ESC) rapid rule-in/rule-out protocols for cTnI results obtained at admission (0h) and 1 hours, as well as 0 h and 2 hours after admission. The rule-out limit will be derived so that the sensitivity and NPV is > 99%, and rule-in limit so that the diagnostic specificity and PPV is > 70% using 60% of the study population. The derived rule-out and rule-in limits will be validated using a remaining population.
Incidence of AEs, ADEs and DDs | Day of admission
  Assess the safety of the SpinChip Platform, as measured by adverse events (AEs), adverse device effects (ADEs) and device deficiencies (DDs).

CONTACTS AND LOCATIONS:
Overall Officials: Helge Røsjø, MD/Professor, Principal Investigator — Akershus University Hospital, Akershus Clinical Research Center (ACR), Norway; Christian Müller, MD/Professor, Principal Investigator — Cardiovascular Research Institute Basel, Switzerland
Locations (9):
- Aarhus Universitetshospital, Aarhus, Denmark
- Universitätsmedizin Göttingen (University Medical Center Göttingen), Göttingen, Germany
- Norway (2):
  - Akershus University hospital, Akershus Clinical Research Center (ACR), Lørenskog, Akerhus
  - Haukland University Hospital, Department of Heart Disease, Bergen, Vestland
- Danderyd University Hospital, Danderyd, Sweden
- Switzerland (2):
  - University hospital Basel, Cardiovascular Research Institute of Basel (CRIB), Basel, Basel
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Alexandra Hospital, Paisley

IPD SHARING:
Plan to Share IPD: No